CLINICAL TRIAL: NCT04276181
Title: Combined Nerve and Tendon Transfer for the Restoration of Hand Function in Individuals With Tetraplegia
Acronym: [CNaTT]
Status: Recruiting | Type: Observational
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Lina Bunketorp Kall, Principal Investigator, Göteborg University
Other Study IDs: 2020-06208; 2020-06208 (Other Grant/Funding Number: The Swedish Research Council); ALFGBG-918931 (Other Grant/Funding Number: The Swedish state under the agreement between the Swedish..); ALFGBG-774951 (Other Grant/Funding Number: The Swedish state under the agreement between the Swedish..)
Record Dates: First submitted 2020-02-07; First posted 2020-02-19 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Spinal Cord Injury Cervical; Tendon Transfer; Nerve Transfer; Rehabilitation; Grip Function

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Combined Nerve and Tendon Transfer (CNaTT) group: The surgical procedures are described in the section Detailed description
- Traditional transfer procedure group: The surgical procedures are described in the section Detailed description

SUMMARY:
Tetraplegia after a cervical spinal cord injury (C-SCI) radically alters an individual's ability to perform normal activities of daily life due to paralysis in all extremities, resulting in lifelong dependence.[1] Traditional tendon transfer surgery has proven successful in restoring grip functions which greatly improves autonomy, but with a restricted passive opening of the hand. The number of transferrable muscles in the arm is however limited, why nerve transfer surgery is a new attractive option to further improve hand function by enabling active opening of the hand. Significant advantages of distal nerve transfers include less extensive surgical dissection, greatly reduced hospital stay, rehabilitation and restrictions, and thereby less health care use and costs. In an effort to further improve hand function and independence in patients with tetraplegia, hand surgeons at Centre for Advanced Reconstruction of Extremities (C.A.R.E.), Sahlgrenska University Hospital (SUH)/Mölndal have developed a strategy in which a nerve transfer procedure aiming to restore active opening of the hand is done prior to reconstruction of grip functions. To date, no study has compared the efficacy of this combined nerve and tendon transfer (CNaTT) procedure to traditional grip reconstruction by means of tendon transfer alone, thus constituting a major gap in the literature. The purpose of this study is therefore to fill that knowledge gap by comparing the clinical outcomes of a cohort of patients who undergo the CNaTT procedure to restore hand function, to those treated by means of tendon transfer alone.

DETAILED DESCRIPTION:
Despite its incurability, surgical reconstruction of arm and hand function is a powerful tool to restore upper limb functions, as well as independence and control in individuals with tetraplegia. Patients with tetraplegia rank better use of the upper limb as their top functional priority, and surgical rehabilitation of the upper limb is proven highly rewarding. Starting in the 70s, pioneering work by dr. Moberg, and continued work by professor Fridén at SUH has guided the development of reconstructive surgical procedures in tetraplegia. As one of the leading units in the field C.A.R.E., SUH/Mölndal is responsible to continue the refinement of surgical treatment strategies. The center works in a value-based patient-oriented environment, with high demands on quality.

The traditional approach to surgical reconstruction of hand function in SCI uses tendon transfer, in which a functionally intact muscle is detached, rerouted and re-attached to a nonworking muscle to replace its original function. By this procedure, finger- and thumb flexion can be successfully and predictably restored, enabling strong active grip functions, but with passive and limited hand opening. Successful nerve transfer surgery in brachial plexus injuries has inspired interest in nerve transfers for patients with C-SCIs. Nerve transfers are conceptually quite similar to tendon transfers but are rarely applied in tetraplegia. To maximize outcome, nerve transfers must be done no later than 1 year after injury. In this procedure, a healthy nerve serving one function is cut and reconnected to a nonfunctional nerve (below the injury level), serving a more important function. Within 6-12 months, the recipient muscle has begun to receive nerve impulses. The preliminary results are very promising and show re-innervation of paralyzed muscles, enabling active opening of the hand. It is an attractive surgical procedure since it allows direct reanimation of the muscle, which is anatomically and mechanically designed to perform that function.

Further advantages of nerve transfers include less extensive surgical dissection, minimal hospital stay, rehabilitation and restrictions, and thereby less health care use and costs. Although the utility of nerve transfers in tetraplegia has yet to be fully determined, early results show promise.

The application of nerve transfer surgery to incomplete tetraplegia offers novel and exciting reconstructive possibilities when combined with tendon transfer techniques, especially in groups with very limited resources. Due to nerve regeneration factors, nerve transfers are not as reliable as tendon transfers, why restoring finger flexion in terms of strength is preferably performed with tendon transfers. It has been suggested that research should be directed at evaluating combined tendon and specific nerve transfer techniques, such as the Bertelli S-PIN (supinator to posterior interosseous nerve transfer) procedure. The S-PIN nerve transfer procedure can reanimate not only the finger extensors, but also allows independent thumb extension and abduction, and thereby enables active opening of the hand. Opening of the hand does not require much strength, and partial outcomes may work satisfactory. The S-PIN procedure combined with the tendon transfer technique has the unique potential to restore hand function to a level as near normal as possible in patients with tetraplegia. This strategy referred to as Combined Nerve and Tendon Transfer (CNaTT) procedure thus allows both opening and strong active closing of the hand, and most likely also result in fewer compensatory movements, which reduces the risk for shoulder pain that interfere with daily activities. At C.A.R.E. there is empirical evidence that support the potential of the combined procedure, such as patients' satisfaction and reporting of being able to better engage in activities in daily life that requires active opening of the hand.

The study has an observational controlled design to which the investigators plan to include 40 cases of CNaTT. As control, patients who undergo tendon transfer alone will be included (due to lack of the prerequisite for nerve transfer; >12 months since injury), in parallel with the cohort of patients who have undergone the traditional procedure in the past (20 prospective cases and 100 historical cases). The results at one year after the tendon transfer procedure will constitute the main outcome.

SURGICAL PROCEDURES

Nerve transfer to achieve opening of the hand by means of Bertelli S-PIN

In this procedure performed bilaterally, the supinator motor nerve gets transferred to the posterior interosseous nerve (S-PIN) according to the technique described by Bertelli. Preoperatively, both donor and recipients nerves and muscles are assessed with electromyography to make sure they are stimulatable on both sides. After a short immobilization period of 2 weeks in a hinged orthosis restricting full extension of the elbow, patients are free to move and train without restrictions. When the first evidence of re-innervation is noticed, patients are instructed to enhancing strength in extensor muscles. Initially, patients activate the donor nerve movement (supination) while the forearm is locked in pronation to facilitate thumb- and finger extension.

The traditional approach to surgical reconstruction of grip by means of tendon transfer

The so-called grip reconstruction is a combination of surgical procedures, customized according to the patient´s needs that can be done many years after a C-SCI. The procedure is developed at SUH by professor Fridén, and has been entitled the alphabet or ABCDEFG procedure, an abbreviation for Advanced Balanced Combined Digital Extensor Flexor Grip reconstruction. The procedure is a one-stage grip and release procedure, a result from several previous studies to improve strength of tendon attachments, early active mobilization etc. The active tendon transfers will typically include brachioradialis to flexor pollicis longus (BR-FPL) transfer and extensor carpi radialis longus to flexor digitorium profundus (ECRL-FDP) transfer. The balancing procedures differ depending on the muscle strength (MRC) after the nerve transfer procedure. A typical OCu 4 patient with some finger extension will undergo: split flexor pollicis longus (FPL)- extensor pollicis longus (EPL) tenodesis, passive reconstruction of the interossei, carpometacarpal (CMC) joint capsulodesis, EPL tenodesis and extensor digiti minimi (EDM)- abductor pollicis brevis (APB) transfer/tenodesis. Our specific and active rehabilitation protocol start within 24 hours after surgery and has previously been described in detail.

ELIGIBILITY:
Inclusion criteria:

* Subjects must be between 15-55 years of age
* Subjects must be diagnosed with a spinal cord injury AIS level C5 to C7
* Time after injury ≤ 12 months
* The strength of the muscle supplied by the donor nerve (supinator) must be graded ≥ 4 according to Medical Research Council (MRC)
* The strength of musculus brachioradialis and wrist extensors must be graded ≥ 4 according to MRC (to be used in grip reconstruction)

Exclusion criteria:

* Finger extensor strength ≤ MRC 1
* Evidence of lower motor neuron injury in muscles supplied by the donor nerve
* Subjects must not have any current serious or unstable illness that could interfere with the study
* Medically unstable to undergo surgery as determined by physician
* Spasticity in the forearm or hand graded > 1 according to Modified Ashworth Scale

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with tetraplegia due to a cervical spinal cord injury.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2020-01-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cylinder test | 5 minutes
  This test is developed at SUH and currently under reliability testing. The cylinder test assesses the patients' ability to actively grasp and release glass cylinders of varying breadth, ranging from 10 to 150 mm.

SECONDARY OUTCOMES:
Grip ability as measured using the Grasp and Release Test (GRT) | 20 minutes
  GRT assesses the ability to pick up, move, and release six objects of varying sizes, weights and textures using a palmar or lateral grasp. Each object represents one or more objects routinely manipulated for activities of daily living (ADL) that represented a range of difficulties.
Grip strength will be measured with JAMAR dynamometer | 2 minutes
Pinch grip strength will be assessed using the Pinch Gauge | 2 minutes
Activity and participation (goal achievement and quality of life) will be measured using the Canadian Occupational Performance Measure (COPM) | 10 minutes
Activity and participation will be measured using the Tetraplegic Upper Limb Activity Questionnaire (TUAQ). | 10 minutes
  Ranges between 13 to 130. Lower scores indicate a higher level of independence.
Satisfaction with surgery will be measured using the Swedish tetraplegia surgery satisfaction questionnaire. | 10 minutes
  Ranges between 20 - 100. Higher scores indicate a higher level of satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Advanced Reconstruction of Extremities, Sahlgrenska University Hospital/Mölndal, Mölndal, Sweden

REFERENCES:
- [Background] Friden J, Gohritz A. Tetraplegia Management Update. J Hand Surg Am. 2015 Dec;40(12):2489-500. doi: 10.1016/j.jhsa.2015.06.003. PMID 26537454
- [Background] Bunketorp-Kall L, Wangdell J, Reinholdt C, Friden J. Satisfaction with upper limb reconstructive surgery in individuals with tetraplegia: the development and reliability of a Swedish self-reported satisfaction questionnaire. Spinal Cord. 2017 Jul;55(7):664-671. doi: 10.1038/sc.2017.12. Epub 2017 Feb 21. PMID 28220821
- [Background] Snoek GJ, IJzerman MJ, Hermens HJ, Maxwell D, Biering-Sorensen F. Survey of the needs of patients with spinal cord injury: impact and priority for improvement in hand function in tetraplegics. Spinal Cord. 2004 Sep;42(9):526-32. doi: 10.1038/sj.sc.3101638. PMID 15224087
- [Background] Moberg E. The present state of surgical rehabilitation of the upper limb in tetraplegia. Paraplegia. 1987 Aug;25(4):351-6. doi: 10.1038/sc.1987.63. No abstract available. PMID 3627823
- [Background] Bossuyt FM, Arnet U, Brinkhof MWG, Eriks-Hoogland I, Lay V, Muller R, Sunnaker M, Hinrichs T; SwiSCI study group. Shoulder pain in the Swiss spinal cord injury community: prevalence and associated factors. Disabil Rehabil. 2018 Apr;40(7):798-805. doi: 10.1080/09638288.2016.1276974. Epub 2017 Jan 13. PMID 28084832
- [Background] van Zyl N, Hahn JB, Cooper CA, Weymouth MD, Flood SJ, Galea MP. Upper limb reinnervation in C6 tetraplegia using a triple nerve transfer: case report. J Hand Surg Am. 2014 Sep;39(9):1779-83. doi: 10.1016/j.jhsa.2014.06.017. Epub 2014 Jul 23. PMID 25063391
- [Background] O'Grady KM, Power HA, Olson JL, Morhart MJ, Harrop AR, Watt MJ, Chan KM. Comparing the Efficacy of Triple Nerve Transfers with Nerve Graft Reconstruction in Upper Trunk Obstetric Brachial Plexus Injury. Plast Reconstr Surg. 2017 Oct;140(4):747-756. doi: 10.1097/PRS.0000000000003668. PMID 28609352
- [Background] Fox IK, Davidge KM, Novak CB, Hoben G, Kahn LC, Juknis N, Ruvinskaya R, Mackinnon SE. Use of peripheral nerve transfers in tetraplegia: evaluation of feasibility and morbidity. Hand (N Y). 2015 Mar;10(1):60-7. doi: 10.1007/s11552-014-9677-z. PMID 25767422
- [Background] Bertelli JA, Ghizoni MF. Nerve transfers for elbow and finger extension reconstruction in midcervical spinal cord injuries. J Neurosurg. 2015 Jan;122(1):121-7. doi: 10.3171/2014.8.JNS14277. PMID 25343189
- [Background] Friden J, Lieber RL. Reach out and grasp the opportunity: reconstructive hand surgery in tetraplegia. J Hand Surg Eur Vol. 2019 May;44(4):343-353. doi: 10.1177/1753193419827814. Epub 2019 Feb 11. PMID 30744461
- [Background] Bertelli JA, Tacca CP, Ghizoni MF, Kechele PR, Santos MA. Transfer of supinator motor branches to the posterior interosseous nerve to reconstruct thumb and finger extension in tetraplegia: case report. J Hand Surg Am. 2010 Oct;35(10):1647-51. doi: 10.1016/j.jhsa.2010.07.012. PMID 20888500
- [Background] Friden J, Reinholdt C, Turcsanyii I, Gohritz A. A single-stage operation for reconstruction of hand flexion, extension, and intrinsic function in tetraplegia: the alphabet procedure. Tech Hand Up Extrem Surg. 2011 Dec;15(4):230-5. doi: 10.1097/BTH.0b013e31821b5896. PMID 22105635
- [Background] Wangdell J, Bunketorp-Kall L, Koch-Borner S, Friden J. Early Active Rehabilitation After Grip Reconstructive Surgery in Tetraplegia. Arch Phys Med Rehabil. 2016 Jun;97(6 Suppl):S117-25. doi: 10.1016/j.apmr.2015.09.025. PMID 27233586